CLINICAL TRIAL: NCT06348615
Title: Sponsored Interventional Single-center Study for the Assessment of the Efficacy and Tolerability of a Medical Device in Crema-gel for the Treatment of PEF (Edemato-fibrosclerotic Panniculopathy of 2nd and 3rd Degree)
Brief Title: Study Aimed at Evaluation of the Effectiveness and Tolerability of an Anti-cellulite Cream Medical Device
Acronym: DEFBODY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ICIM International S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEFBODY
Record Dates: First submitted 2024-01-25; First posted 2024-04-05 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cellulite
Keywords: cellulite; anti-cellulite treatment; 2nd and 3rd degree cellulite; medical device for the treatment of cellulite; cream-gel for cellulite; edematous fibrosclerotic panniculopathy
MeSH Terms: conditions — Cellulite; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: 1 bottle (cream-gel) 400ml (Experimental): Each study subject applies the medical device (one cream-gel of 400ml) on both buttocks and thighs affected by cellulite (II or III degree) massaging with circular movements following the direction of the lymphatic flow, twice a day for 4 weeks ( intermediate visit) and for another 8 weeks (final visit).
  If the device is finished during the study, a new device may be provided, always one cream-gel of 400 ml.
  Interventions: Device: Anti-cellulite cream-gel Medical Device (DEFBODY)

INTERVENTIONS:
Device: Anti-cellulite cream-gel Medical Device (DEFBODY) — one bottle of 400 ml, twice a day

SUMMARY:
Post-marketing clinical study conducted on a CE medical device, named Defense Body, cellulite treatment, edematous fibrosclerotic panniculopathy (2nd and 3rd stage pathology), reducing draining cream-gel, to verify its effectiveness and tolerability on a panel of 56 subjects females affected by 2nd and 3rd degree PEF. The effectiveness of the device is measured in terms of reduction in thigh circumference, improvement in the appearance of the skin with reduction of the orange peel appearance and improvement in skin smoothness.

DETAILED DESCRIPTION:
Post-marketing, sponsored, interventional, single-centre clinical study conducted on a medical device, already CE marked, named Defense Body cellulite treatment edematous fibrosclerotic panniculopathy (2nd and 3rd stage pathology) draining reducing gel-cream, to verify the its efficacy and tolerability on a panel of 56 female subjects, aged between 18 and 55, in good general health, and suffering from 2nd and 3rd degree PEF.

A comparison study will be carried out between the clinical condition of the subjects at baseline T0, compared to the condition at the end of treatment T2, with provision for an intermediate visit halfway through treatment, T1.

At the first enrollment visit (T0), the patient will be subjected to anthropometric measurements, measurement of the skin profile of the thigh, measurement of the thigh circumference and evaluation by the clinician of the degree of cellulite using pinch tests and digital photographs of the area. treated in profile and three-quarter view.

After 4 (± 3 days) (T1) and 8 weeks (± 4 days) (T2) from the start of the study, the patient is visited again.

The Doctor will repeat the assessments described at T0, with the addition of verifying continued compliance with the enrollment criteria; overall evaluation by the patient of satisfaction and compliance; recording of each AE or AED or drop-off; recording of any concomitant pharmacological treatment.

The patient's overall assessment of satisfaction and compliance will be carried out only at the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Age between 18 and 55;
* Presence of grade II or III symmetrical cellulite on the right and left lower limbs;
* BMI between 18.5 and 30;
* Good state of health and absence of chronic pathologies;
* Willingness not to change one's lifestyle during study;
* Willingness to join the study and sign the information consent.

Exclusion Criteria:

* Subjects being treated with other topical products in the lower limbs;
* Subjects being treated with other topical or systemic cellulite products;
* Subjects with skin conditions and/or inflammatory conditions underway or had in the period immediately preceding the start of the study;
* Subjects with a history of venous or lymphatic insufficiency in the lower limbs;
* Subjects with known allergies or intolerances to one of the components of the product;
* Pregnant or breastfeeding subjects;
* Subjects undergoing slimming therapy, whether pharmacological or dietary;
* Subjects who practice intense or competitive sporting activity.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
First day of study initiation: clinical history; personal and demographic data and previous or concomitant treatments | First day: within 24 hours
  The following activities are planned on the first day:
  * clinical history of the recruited subjects;
  * personal and demographic data;
  * previous and/or concomitant treatments.
First day of study initiation: BMI | First day: within 24 hours
  Evaluation of height (cm) and weight (Kg) for the calculation of the body mass index, considered in the range 18.5 - 30.
First day of study initiation: Measurement of waist circumference, hip circumference and thigh circumference | First day: within 24 hours
  Measurement of:
  * waist circumference;
  * hip circumference
  * thigh circumference
  These measurements are taken using a flexible tape measure with the subject barefoot, in an upright position and, in the specific case of the measurement of the thigh, 1 cm below the crease of the buttock.
First day of study initiation: digital photographs of the area to be treated | First day: within 24 hours
  digital photographs of the area to be treated, taken in profile and three-quarter view with a model camera Nikon Digital Camera.
First day of study initiation: skin profilemetry of the thigh | First day: within 24 hours
  Evaluation of the skin profilemetry of the thigh in a predetermined target area, through a computerized analysis Antera 3D CS Camera and 3.X software set (Mitavex, Dublin, Ireland).
  The images obtained allow the operator to measure the volume of protrusion and skin depressions in the area, expressed in mm3.
First day of study initiation: pinch test | First day: within 24 hours
  The clinician evaluates the degree of cellulite using a pinch test by applying pressure on the skin between thumb and index finger and assigns a grade from 0 to 4 according to a specific table.

SECONDARY OUTCOMES:
After 28 days of treatment: recording of any concomitant pharmacological treatments that have occurred. | On the 28th day of treatment
  Any concomitant pharmacological treatments that have occurred are evaluated and recorded.
After 28 days of treatment: BMI | On the 28th day of treatment
  Evaluation of height (cm) and weight (Kg) for the calculation of the body mass index, considered in the range 18.5 - 30.
  In particular, at T2 the minimum acceptable clinical improvement in skin profile measurement will be evaluated (equal to a reduction in the depth of skin depressions of 8-10 mm3.
After 28 days of treatment: Measurement of waist circumference, hip circumference and thigh circumference | On the 28th day of treatment
  Measurement of:
  * waist circumference;
  * hip circumference;
  * thigh circumference.
  These measurements are taken using a flexible tape measure with the subject barefoot, in an upright position and, in the specific case of the measurement of the thigh, 1 cm below the crease of the buttock.
After 28 days of treatment: digital photographs of the area to be treated | On the 28th day of treatment
  Digital photographs of the area to be treated, taken in profile and three-quarter view with a model camera Nikon Digital Camera.
After 28 days of treatment: skin profilemetry of the thigh | On the 28th day of treatment
  Evaluation of the skin profilemetry of the thigh in a predetermined target area, through a computerized analysis Antera 3D CS Camera and 3.X software set (Mitavex, Dublin, Ireland).
  The images obtained allow the operator to measure the volume of protrusion and skin depressions in the area, expressed in mm3.
After 28 days of treatment: pinch test | On the 28th day of treatment
  The clinician evaluates the degree of cellulite using a pinch test by applying pressure on the skin between thumb and index finger and assigns a grade from 0 to 4 according to a specific table.
After 28 days of treatment: AE or AED or Drop-off | On the 28th day of treatment
  Recording of any adverse event (AE) or adverse device event (AED) or drop-off.
After 28 days of treatment: satisfaction evaluation and compliance | On the 28th day of treatment
  Overall evaluation by each clinical study subject of satisfaction and compliance.
After 56 days of treatment: recording of any concomitant pharmacological treatments that have occurred. | On the 56th day of treatment
  Any concomitant pharmacological treatments that have occurred are evaluated and recorded.
After 56 days of treatment: BMI | On the 56th day of treatment
  Evaluation of height (cm) and weight (Kg) for the calculation of the body mass index, considered in the range 18.5 - 30.
  In particular, at T2 the minimum acceptable clinical improvement in skin profile measurement will be evaluated (equal to a reduction in the depth of skin depressions of 8-10 mm3.
After 56 days of treatment: Measurement of waist circumference, hip circumference and thigh circumference | On the 56th day of treatment
  Measurement of:
  * waist circumference;
  * hip circumference;
  * thigh circumference.
  These measurements are taken using a flexible tape measure with the subject barefoot, in an upright position and, in the specific case of the measurement of the thigh, 1 cm below the crease of the buttock.
After 56 days of treatment: digital photographs of the area to be treated | On the 56th day of treatment
  Digital photographs of the area to be treated, taken in profile and three-quarter view with a model camera Nikon Digital Camera.
After 56 days of treatment: skin profilemetry of the thigh | On the 56th day of treatment
  Evaluation of the skin profilemetry of the thigh in a predetermined target area, through a computerized analysis Antera 3D CS Camera and 3.X software set (Mitavex, Dublin, Ireland).
  The images obtained allow the operator to measure the volume of protrusion and skin depressions in the area, expressed in mm3.
After 56 days of treatment: pinch test | On the 56th day of treatment
  The images obtained allow the operator to measure the volume of protrusion and skin depressions in the area, expressed in mm3.
After 56 days of treatment: AE or AED or Drop-off | On the 56th day of treatment
  Recording of any adverse event (AE) or adverse device event (AED) or drop-off.
After 56 days of treatment: evaluation of compliance | On the 56th day of treatment
  Evaluation of compliance by each clinical study subject.
  Adherence to the treatment is verified by asking the patient to keep a diary in which to note the morning and evening application, any adverse events that may occur and any medication taken.
After 56 days of treatment: overall rating of product satisfaction | On the 56th day of treatment
  For the overall evaluation of patient satisfaction with the product, subjects will be asked to respond to a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Santo Raffaele Mercuri, Principal Investigator — I.R.C.C.S. Ospedale San Raffaele
Locations (1):
- Dermatology Unit - I.R.C.C.S. Ospedale San Raffaele, Milan, Italy